CLINICAL TRIAL: NCT06267586
Title: Examining the Effects of PeptiSleep, a Plant-based Sleep Aid, in Healthy Males and Females With Mild to Moderate Sleep Impairment
Brief Title: Effects of PeptiSleep in Healthy Males and Females With Mild to Moderate Sleep Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Collaborators: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PN23.007
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Randomized, single-blind, placebo-controlled, parallel dose response study conducted over 70 days
Who Masked: Participant
Masking Description: Participants will be unaware of arm allocation however as each arm contains a different number of capsules to be consumed, the investigator will be aware of the arm allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- PeptiSleep 250 mg/day (Experimental): Low dose Given as 1 capsule 1 hour before bed
  Interventions: Dietary Supplement: PeptiSleep
- PeptiSleep 500 mg/day (Experimental): Middle dose Given as 2 capsules 1 hour before bed
  Interventions: Dietary Supplement: PeptiSleep
- PeptiSleep 1000 mg/day (Experimental): High dose Given as 4 capsules 1 hour before bed
  Interventions: Dietary Supplement: PeptiSleep
- Microcrystalline Cellulose 500mg/day (Placebo Comparator): Placebo Given as 2 capsules 1 hour before bed
  Interventions: Dietary Supplement: Placebo MCC micro-crystalline cellulose

INTERVENTIONS:
Dietary Supplement: PeptiSleep — Plant protein hydrolysate
  Arms: PeptiSleep 1000 mg/day; PeptiSleep 250 mg/day; PeptiSleep 500 mg/day
Dietary Supplement: Placebo MCC micro-crystalline cellulose — Placebo MCC micro-crystalline cellulose
  Arms: Microcrystalline Cellulose 500mg/day

SUMMARY:
Examining the effects of PeptiSleep, a plant-based sleep aid, in healthy males and females with mild to moderate sleep impairment

DETAILED DESCRIPTION:
The primary aim of this is a first in human study is to evaluate safety and establish the effective dose in males and females who experience mild to moderate sleep impairment, but who are otherwise healthy. PeptiSleep will be supplemented one hour before bed as a single oral dose of either 250mg, 500mg or 1000mg/day. A placebo group will also be included who will receive 500mg of microcrystalline cellulose.

This trial incorporates a sleep tracking element to measure sleep quality and quantity via a ring which will be worn by participants for the duration of the study. The trial will be conducted over 10 weeks, which includes a 2 week run-in period to gather baseline sleep data, followed by 8 weeks of PeptiSleep supplementation and sleep tracking.

The primary endpoint will measure safety and tolerability via adverse event reporting and incidence rate ratio between placebo and PeptiSleep from baseline to the end of the study period.

Secondary endpoints investigated during the trial will include changes sleep quantity and quality, insomnia severity, daytime sleepiness, stress and anxiety, alertness, and biochemistry markers (melatonin, serotonin, CRP, TNFα, IL-6, E/LFT).

Exploratory endpoints will include various sleep metrics measured via the wearable tracker including heart rate variability, sleep efficiency, respiratory rate, blood oxygen sensing and daily readiness score.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18-65 years
* Generally healthy
* BMI 18.5 - 33.0.kg/m2
* Volunteers who score 0-14 on the ISI screening questionnaire (to exclude insomniacs)
* Those with an average sleep score of 89 or less as determined by the sleep tracker during the 14-day run-in period
* Must be willing to wear the sleep tracker for the duration of their enrolment
* Able to provide informed consent
* Agree not to change current diet and/or exercise frequency or intensity during entire enrolment period
* Agree not to use other medicines or supplements for sleep, stress, depression, or anxiety other than the test product during enrolment period
* Agree to not participate in another clinical trial during enrolment period

Exclusion Criteria:

* Those diagnosed with a chronic sleep disorder, insomnia, restless leg syndrome, sleep apnoea or score of 15 or more on ISI questionnaire
* Those with an average sleep score of 90 or over as determined by the sleep tracker during the 14-day run-in period
* Those deemed unsuitable based on data from the sleep tracker measurements collected during the 14-day run in period i.e., those with non-wear time exceeding a 24-hour period on more than one occasion
* Those using medications which induce CYP3A4 such as phenobarbital, phenytoin, rifampicin, St. John's Wort, and glucocorticoids.
* Those using prescription or OTC medications or supplements for sleep, stress, depression or anxiety including CBD within 1 month prior to enrolment.
* Those using aromatherapy to help manage sleep, stress, depression, or anxiety within 1 month prior to enrolment.
* Use of a digital device (besides the supplied sleep tracker) to help monitor or manage sleep during the study period.
* Current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Serious illness1 e.g., mood disorders such as depression, anxiety or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease or heart conditions
* Unstable illness2 e.g., diabetes and thyroid gland dysfunction
* Diagnosed or consistent gastrointestinal issues that disrupt sleep.
* History of renal function impairment
* Volunteers with COPD or a chronic breathing disorder
* Currently taking Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin or other anticoagulation therapy including low dose aspirin
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Regularly taking stimulants (e.g., coffee, caffeine supplements, beverages containing caffeine) 5 hours before bed
* Regularly consuming more than 500mg of caffeine per day
* Those working night-shift employment who are unable to have a normal night's sleep.
* Disturbed sleeping pattern caused by external factors (e.g., young children, partner etc.)
* Pregnant or lactating women
* Allergic, sensitive, or intolerant to any of the ingredients in active or placebo formula
* Participants who are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 1 month and any other sleep clinical trial during the past 3 months.
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion.

  1. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.
  2. An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of a dose range of PeptiSleep via adverse event reporting | Day 0 to 56
  Change from baseline to the end of the study period in safety via adverse event reporting and incident rate ratio between placebo and a dose range of PeptiSleep

SECONDARY OUTCOMES:
Safety via electrolytes and liver function tests | Day 0 to 56
  Change from baseline to the end of the study period in safety including electrolytes and liver function markers via blood test
Sleep Quality via Leeds Sleep Evaluation Questionnaire | Day 0 to 56
  Change from baseline to the end of the study period in Sleep Quality via Leeds Sleep Evaluation Questionnaire (LSEQ). The LSEQ comprises ten self-rating 100-mm-line analogue questions concerned with aspects of sleep and early morning behaviour. A visual analogue scale is used with two extreme states defined at the ends of the line (e. g. Tired = score of 0, Alert = score of 10). The subject responds by placing a vertical mark on the line to indicate his present self- evaluation.
  The four subscales are as follows:
  * The ease of getting to sleep (GTS), questions 1-3
  * The perceived quality of sleep (QOS), questions 4-5
  * The easy of awakening from sleep (AFS), questions 6-7
  * The integrity of behaviour following wakefulness (BFW), questions, 8-10
Insomnia severity via the Insomnia Severity Index Questionnaire | Day 0 to 56
  Change from baseline to the end of the study period in Insomnia Severity via Insomnia Severity Index (ISI). The questionnaire has seven questions. The seven answers are added up to get a total score.
  Total score categories:
  * 0-7 = No clinically significant insomnia
  * 8-14 = Subthreshold insomnia
  * 15-21 = Clinical insomnia (moderate severity)
  * 22-28 = Clinical insomnia (severe)
Sleep onset time via self-reported recording in a Sleep Diary | Day 0 to 56
  Change from baseline to the end of the study period in Sleep Onset Time via Consensus Sleep Diary (CSD)
Sleep pattern via self-reported recording in a Sleep Diary | Day 0 to 56
  Change from baseline to the end of the study period in self reported Sleeping Pattern and number of Disturbance as recorded using a Consensus Sleep Diary (CSD)
Daytime Sleepiness via the Epworth Sleepiness Scale | Day 0 to 56
  Change from baseline to the end of the study period in Day Time Sleepiness and Nap Count via the Epworth Sleepiness Scale (ESS). The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher the propensity for daytime sleepiness
  * Scores 0-5 Lower Normal Daytime Sleepiness
  * Scores 6-10 Higher Normal Daytime Sleepiness
  * Scores 11-12 Mild Excessive Daytime Sleepiness
  * Scores 13-15 Moderate Excessive Daytime Sleepiness
  * Scores 16-24 Severe Excessive Daytime Sleepiness.
Stress via the Perceived Stress Scale | Day 0 to 56
  Change from baseline to the end of the study period in Stress via a self reported questionnaire - Perceived Stress Scale (PSS). The questions in this scale ask about feelings and thoughts during the last month. The questionnaire asks the participant to indicate how often they felt or thought a certain way with 0 meaning never and 4 meaning very often.
  PSS scores are calculated by:
  * First, reverse your scores for questions 4, 5, 7, and 8. On these 4 questions, change the scores like this: 0 = 4, 1 = 3, 2 = 2, 3 = 1, 4 = 0.
  * Add up your scores for each item to get a total.
  * Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
    * Scores ranging from 0-13 would be considered low stress.
    * Scores ranging from 14-26 would be considered moderate stress.
    * Scores ranging from 27-40 would be considered high perceived stress
Stress via self reported Profile of Mood States Questionnaire | Day 0 to 56
  Change from baseline to the end of the study period in Stress via a self reported questionnaire called Profile of Mood States (POMS). The questionnaire contains 65 words that describe feelings which are rated from 0-4. Scores are calculated:
  * Tension = Tense, Shaky, On Edge, Panicky, Relaxed, Uneasy, Restless, Nervous and Anxious
  * Depression = Unhappy, Sorry for Things Done, Sad, Blue, Hopeless, Unworthy, Discouraged, Lonely, Miserable, Gloomy, Desperate, Helpless, Worthless, Terrified and Guilty
  * Anger = Anger, Peeved, Grouchy, Spiteful, Annoyed, Resentful, Bitter, Ready to Fight, Rebellious, Deceived, Furious and Bad Tempered
  * Fatigue = Worn Out, Listless, Fatigued, Exhausted, Sluggish, Weary and Bushed
  * Confusion= Confused, Unable to Concentrate, Muddled, Bewildered, Efficient, Forgetful, and Uncertain About Things
  * Vigour =Lively, Active, Energetic, Cheerful, Alert, Full of Pep, Carefree and Vigorous
Anxiety via self-reported Beck Anxiety Inventory questionnaire | Day 0 to 56
  Change from baseline to the end of the study period in Anxiety via Beck Anxiety Inventory (BAI) questionnaire. The BAI consists of 21 self-reported items on a four-point scale - ''not at all'' (0) to ''severely'' (3) to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63
  * Minimal anxiety levels (0-7)
  * Mild anxiety (8-15)
  * Moderate anxiety (16-25)
  * Severe anxiety (26-63)
Stress via Salivary cortisol test | Day 0 to 56
  Change from baseline to the end of the study period in Stress via Salivary cortisol test
Alertness via Reaction Time Test | Day 0 to 56
  Change from baseline to the end of the study period in Alertness via Reaction Time Test
Circadian cycles via melatonin and serotonin via blood test | Day 0 to 56
  Change from baseline to the end of the study period in markers associated with circadian cycles - melatonin and serotonin via blood test
Markers associated with inflammation via blood test | Day 0 to 56
  Change from baseline to the end of the study period in Inflammatory Markers such as CRP, TNF-α and IL-6 via blood test
Sleep onset latency via wearable sleep tracker | Day 0 to 56
  Change from baseline to the end of the study sleep onset latency measured in minutes using a wearable sleep tracker
Total sleep time spent in sleep phases via wearable sleep tracker | Day 0 to 56
  Change from baseline to the end of the study in total sleep time during phases of light, deep and REM sleep measured in minutes via a wearable sleep tracker
Blood pressure via blood pressure machine | Day 0 to 56
  Change from baseline to the end of the study in blood pressure measured in mmHG
Heart rate via blood pressure machine | Day 0 to 56
  Change from baseline to the end of the study in heart rate measured in beats per minute using a blood pressure machine
Body Temperature via wearable sleep tracker | Day 0 to 56
  Change from baseline to the end of the study in body temperature measured in Celsius using a wearable sleep tracker
BMI via height and weight measurements | Day 0 to 56
  Change from baseline to the end of the study in BMI. The BMI is calculated by dividing weight in kilograms by height in meters squared and is measured in kg/m2.

OTHER OUTCOMES:
Bedtime via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Bedtime as an estimate of initial period intending to sleep as measured via a wearable sleep tracker
Total time awake via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Total time awake in minutes via a wearable sleep tracker
Sleep quantity via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Sleep quantity measured as the number of hours between bedtime and wake-up time via a wearable sleep tracker
Sleep efficiency via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Sleep efficiency. Sleep efficiency is the percentage of time spent asleep while in bed. It is calculated by dividing the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes). A normal sleep efficiency is considered to be 85% or higher.
Sleep score via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Sleep score Sleep Score ranges 0-100.
  * Scores 85 or higher: Optimal
  * Scores 70-84: Good
  * Under 70: Poor
Nocturnal heart rate via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Nocturnal heart rate, the number of heart beats per minute while at rest via a wearable sleep tracker
Heart Rate variability via wearable sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Heart Rate variability recorded as the time interval between two heartbeats in milliseconds via a wearable sleep tracker
Blood Oxygen sensing via sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Blood Oxygen sensing as measured via the sleep tracking device
Respiratory rate via sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in respiratory rate as measured via the sleep tracking device
Daily Readiness Score via sleep tracker | Day -12 to 0 and Day 0 to 56. Run in period will identify sleep pattern prior to supplementation
  Changes over the course of the study in Daily Readiness Score Readiness Score ranges 0-100.
  * Scores 85 or higher: Optimal
  * Scores 70-84: Good
  * Under 70: Poor

CONTACTS AND LOCATIONS:
Locations (1):
- RDC Clinical, Brisbane, Fortitude Valley Queensland, Australia

IPD SHARING:
Plan to Share IPD: No